CLINICAL TRIAL: NCT07292766
Title: Metabolomic Profiling of Patients With Traumatic Brain Injury
Status: Recruiting | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ekin Guran, MD, Attending anesthesiologist, Aksaray University Training and Research Hospital
Other Study IDs: TBI_omics
Record Dates: First submitted 2025-07-28; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Traumatic Brain Injury; Traumatic Brain Injury (TBI) Patients
Keywords: traumatic brain injury; metabolomics
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — venous blood sample for metabolomic analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TBI: Patients aged 18-65 years with a diagnosis of severe TBI based on clinical or National Institute for Health and Care Excellence (NICE) criteria (post-traumatic imaging)
- Non_TBI: Patients aged 18-65 years who had a traumatic injury without TBI

SUMMARY:
Traumatic Brain Injury (TBI) is a significant cause of mortality and morbidity worldwide. However, the literature on determining its severity and predicting prognosis is insufficient. This study aimed to examine the differences in metabolite levels between trauma patients with severe TBI and orthopedic trauma patients without brain injury.

DETAILED DESCRIPTION:
Traumatic Brain Injury (TBI) is a significant cause of mortality and morbidity worldwide, particularly in young people. TBI is a complex metabolic process associated with an energy crisis resulting from multiple mechanisms, including ischemia, diffusion hypoxia, and mitochondrial dysfunction. Because metabolic derangement is a fundamental component of TBI pathophysiology, these metabolic changes may provide prognostic information and guide treatment. Additionally, the release of brain-specific metabolites (i.e., small molecules with a molecular mass below 500 Da) into the systemic circulation may provide insights into blood-brain barrier (BBB) dysfunction, a fundamental process in TBI. Metabolomic profiling studies are introductory and valuable for elucidating this metabolic process.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65
* Patients diagnosed with severe TBI clinically or according to National Institute for Health and Care Excellence (NICE) criteria (including post-traumatic imaging)
* Patients with non-TBI orthopedic or multitrauma

Exclusion Criteria:

* Presence of brain pathology in the pre-trauma period
* Patient with chronic subdural hematoma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trauma patients with or without TBI, aged between 18 and 65 years, who applied to Aksaray UniversityTraining and Research Hospital will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
metabolomic analysis | Day 1
  Venous blood samples are taken from the participants after the injury. Samples will be analysed using LC/MS. All relevant metabolomes and their respective metabolic pathways will be evaluated using the "KEGG Pathway database".

CONTACTS AND LOCATIONS:
Locations (1):
- Aksaray University, Aksaray, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Banoei MM, Lee CH, Hutchison J, Panenka W, Wellington C, Wishart DS, Winston BW; Canadian biobank, database for Traumatic Brain Injury (CanTBI) investigators, the Canadian Critical Care Translational Biology Group (CCCTBG), the Canadian Traumatic Brain Injury Research, Clinical Network (CTRC). Using metabolomics to predict severe traumatic brain injury outcome (GOSE) at 3 and 12 months. Crit Care. 2023 Jul 22;27(1):295. doi: 10.1186/s13054-023-04573-9. PMID 37481590
- [Result] Zhou M, Liu YW, He YH, Zhang JY, Guo H, Wang H, Ren JK, Su YX, Yang T, Li JB, He WH, Ma PJ, Mi MT, Dai SS. FOXO1 reshapes neutrophils to aggravate acute brain damage and promote late depression after traumatic brain injury. Mil Med Res. 2024 Mar 31;11(1):20. doi: 10.1186/s40779-024-00523-w. PMID 38556884
- [Result] Fedoruk RP, Lee CH, Banoei MM, Winston BW. Metabolomics in severe traumatic brain injury: a scoping review. BMC Neurosci. 2023 Oct 16;24(1):54. doi: 10.1186/s12868-023-00824-1. PMID 37845610